CLINICAL TRIAL: NCT05112211
Title: A Multi-model Image to Evaluate the Efficacy of Doxycycline in Thyroid Associated Ophthalmopathy
Brief Title: Multi-model Image of Doxycycline in TAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, principal investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TAODOXYIMAGE
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-04

CONDITIONS: Thyroid Associated Ophthalmopathy
Keywords: Doxycycline; Thyroid Associated Ophthalmopathy; Extraorbital muscle; Orbit fat volume; Multi-modal image
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Patients diagnosed by Thyroid-Associated Ophthalmopahty
Masking Description: Assessors who calculate the changes of the images are masked of the diagnosis and treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- doxycycline (Experimental): patients administrated with doxycycline tablets 100mg orally per day
  Interventions: Drug: Doxycycline Hyclate

INTERVENTIONS:
Drug: Doxycycline Hyclate — patients administrated with doxycycline tablets 100mg orally per day

SUMMARY:
This study aims to evaluate the efficacy of doxycycline treating Thyroid Associated Ophthalmopathy by multi-modal image.

DETAILED DESCRIPTION:
Thyroid Associated Ophthalmopathy is one of autoimmune orbital diseases characterized by enlargement of the extraocular muscles and increase in fatty or/and orbit connective tissue volume affecting the appearance and visual function of the eyes. Different degrees of exophthalmos, eyelid aperture, lid retraction and lid lag are common symptoms apprearing in TAO. The improvement of exophthalmos is usually measured with Hertel instrument and the change of eyelid is measured with millimeter ruler. All these measurements are subjective, low reliable and less accurate.

TAO can be classified into active phase and inactive phase according to the activity score and wait-and-see or surgery are widely chosen for patients in inactive phase. But still a progression and reoccurrence can be a big challenge for ophthalmologists. This is a perspective cohort study to evaluate the efficacy of doxycycline in TAO by multi-model image.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18-70 years old
* Diagnosed with TAO

Exclusion Criteria:

* Sight-threatening TAO with dysthyroid optic neuropathy
* Allergy of tetracycline
* Have contraindications of MRI(metal pacemaker, fake teeth, foreign body and other materials which will disturb the examination)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
change of extraocular muscle volume and orbital fat volume by MRI | at month 6
  3D MRI image will be established and the volume of extraocular muscle and orbital fat will be calculated by the same advanced programmer who is blinded of the pre- or post- treatment images order. A higher score means a better outcome.

SECONDARY OUTCOMES:
change of exophthalmos | at month 6
  exophthalmos will be measured by the same investigator using the same Hertel instrument.
  A higher change of exphthalmos means a better outcome.
change of Quality of Life | at month 6
  The score of quality of life will be assessed by the same investigator using GO-QoL. The better change of quality of life means a better outcome.
change of eyelid aperture, lid retraction and lid lag | at month 6
  the values will be measured by the same investigator using the same millimeter ruler and the higher values change, the better the outcome is.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No